CLINICAL TRIAL: NCT02260856
Title: PEDS Trial: Percutaneous Epiphysiodesis, Drill Versus Screws for Leg Length Discrepancy a Randomized Clinical Trial
Brief Title: A Randomized Controlled Trial of Leg Length Discrepancy Techniques
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study expired December 16, 2023 and inactivated due to non response to continuing review 2/1/24. Study never reactivated so it was terminated.
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Boston Children's Hospital (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-174
Record Dates: First submitted 2014-06-26; First posted 2014-10-09 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Leg Length Discrepancy
Keywords: RCT; Epiphysiodesis; Tantalum beads; Patient centered outcome data; Cost effective analysis
MeSH Terms: conditions — Leg Length Inequality | interventions — Sterilization, Reproductive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous Drill Epiphysiodesis (Active Comparator): A 5 mm incision will be made centered over the physis both medially and laterally. A 4.5 mm drill will be passed repeatedly across the physis in a divergent manner. Curettes will then be used to further remove and disrupt the growth plate. Fluoroscopy will be used throughout to ensure proper passage of the drill and curettes. Omnipaque dye will then be inserted to confirm ablation of the physis.
  Interventions: Device: Tantalum Beads & Injector; Procedure: Percutaneous Drill Epiphysiodesis
- Percutaneous Screw Epiphysiodesis (Experimental): In the distal femur, guide wires will be placed in an antegrade fashion, with an 8 mm skin incision proximal to the physis both medially and laterally. The guide wire will be placed with the medial wire crossing the physis at the junction of the middle and medial third of the physis. The lateral guide wire will cross the physis at the junction of the lateral and middle third of the physis. The wires will extend into the epiphysis, but will not enter the joint. The guide wires will be over drilled with a 5 mm drill, and 7.3 mm fully threaded cannulated screws will be placed across the growth plate. For tibias, screw placement will be retrograde, with 8 mm incisions made medially and laterally distal to the physis, with guide wires aiming proximally.
  Interventions: Device: Tantalum Beads & Injector; Procedure: Percutaneous Screw Epiphysiodesis

INTERVENTIONS:
Device: Tantalum Beads & Injector — To measure growth at physis, four tantalum beads will be implanted per physis at baseline and take radiostereometric analysis measurements at all follow up timepoints. Tantalum beads have been used to make detailed three dimensional radiographic measurements in orthopedic and other specialties
  Other Names: RSA Biomedical.; One (1) UmRSA® Injectors Conventional design, Mussle loaded; Robust design, Easy to clean and sterilize, Modular design; (for Tantalum Markers diameter 0.8 or1.0mm); 500 RSA ®Tantalum Markers diameter 0.8mm or 1.0mm
Procedure: Percutaneous Drill Epiphysiodesis
  Arms: Percutaneous Drill Epiphysiodesis
Procedure: Percutaneous Screw Epiphysiodesis
  Arms: Percutaneous Screw Epiphysiodesis

SUMMARY:
This is a randomized clinical trial of epiphysiodesis techniques: percutaneous transphyseal screw epiphysiodesis versus percutaneous drill epiphysiodesis for the correction of leg length discrepancy. Failed epiphysiodesis was selected as the primary outcome. Failed epiphysiodesis was defined as one or more of the following: development of angular deformity > 5°, revision epiphysiodesis, or growth inhibition < 70% of expected. EOS, low dose biplanar X-Ray, will be used to make all length measurements. Secondary outcomes assess mean growth at the physis following epiphysiodesis, in the subset of patients with bead implantation, fluoroscopy and operative times, length of stay, return to full weight bearing, as well as functional and quality of life outcomes. The following outcome scales will be used to measure pain (VAS), quality of life (PROMIS Pediatric Pain Interference Scale), and function (PROMIS Pediatric Mobility Scale, Pedi-FABS, and UCLA Activity Score). Each of these scales has been validated for use in children (Beyer, Denyes, & Villarruel, 1992; DeWitt et al., 2011; Fabricant et al., 2013; Novais et al., 2014; Varni et al., 2010a). We will also determine the cost associated with each technique and perform a cost-effectiveness analysis to establish which technique is preferred from a societal perspective.

DETAILED DESCRIPTION:
Drill and screw epiphysiodesis are the two most common techniques for surgical correction of predicted limb length discrepancies 2-5cm. Both procedures require minimal incisions, less than 1cm, (Canale & Christian, 1990; Metaizeau et al., 1998). Previous studies have demonstrated that both drill and screw epiphysiodesis result in improved outcomes compared to open techniques (Alzahrani, Behairy, Alhossan, Arab, & Alammari, 2003; Canale & Christian, 1990). Moreover, alternative approaches such as medial and lateral 8 plates may not sufficiently tether growth, or cause peripheral but not central growth arrest (Stewart et al., 2013). We selected drill vs. screw epiphysiodesis as the two treatment groups as they are both minimally invasive, relatively effective, in common usage, and are thought to differ in costs and other characteristics.

Although outcomes of drill and screw epiphysiodesis exist{{10 Campens,C. 2010; 11 Ghanem,I. 2011}} , the assessments are retrospective non-randomized series, which may be at risk for selection bias, and may not adequately capture all of the outcomes of interest, depending on what data is routinely collected and documented in the medical chart. To our knowledge, no prospective randomized comparison of epiphysiodesis techniques and clinical outcomes has been published accurately assessing how effective each technique is in disabling growth at the physis, or taking into account patient-centered outcomes or cost. Operative measures such as the surgical time and radiation exposure from intra-operative fluoroscopy have not previously been compared. Patient-centered outcomes such as level of pain, activity, and function by measures such PROMIS and Ped-FABS, have not been previously assessed in this population. The proposed research study aims to fill this gap.

This study was designed as a multicenter randomized trial to answer an important clinical question and to do so with a clearly defined objective and validated outcomes. This trial can be executed on a relatively small budget with simple outcome measures, and recruitment of a moderate number of patients at each of a few centers well equipped for research. By involving multiple surgeons and patients from various geographies, we improve the generalizability of this study. Our institution and collaborating institutions have been successful in completing randomized clinical trials in the past. This study will answer a clinical question that is important and current, providing orthopedic surgeons with an evidence-based identification of the ideal technique for treating predicted limb length discrepancies 2-7cm.

This study will also be the first to accurately measure mean growth following both epiphysiodesis techniques, through implantation of tantalum beads in consenting participants. These beads will provide stationary landmarks by which growth can be measured directly, and not inferred. Previous methods of judging epiphysiodesis success have primarily relied on assessing efficacy by estimating growth inhibition through calculation. Tantalum beads have been successfully used in adults and children (Lauge-Pedersen,H. 2006), and although it requires implantation of small radio-opaque beads, it is considered the gold standard when making detailed radiographic measures, and the optimal technique for physeal growth measurements.(Lauge-Pedersen,H. 2006)(Haugan,K. 2012). Over 300 000 beads have been inserted in vivo without significant complications.

ELIGIBILITY:
Inclusion Criteria:

* Open growth plates
* Skeletally immature requiring isolated complete epiphysiodesis of the distal femur and/or proximal tibia
* At least one year of predicted growth remaining
* Less than 18 years of age
* Predicted limb length discrepancy 2-7 cm

Exclusion Criteria:

* Patients undergoing additional orthopedic procedures at time of epiphysiodesis
* Metabolic bone disease or "sick physis" syndrome, that may cause bone to grow in an unpredictable manner.
* Pregnancy

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2015-06; Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Failure of Epiphysiodesis | 2-6 weeks, 5-7 months, 11-13 months, 23-25 months, 59-61 months
  development of angular deformity > 5°, revision epiphysiodesis, or growth inhibition < 70% of expected

SECONDARY OUTCOMES:
Change in Physeal Growth | Baseline, 2-6 weeks, 5-7 months, 11-13 months, 23-25 months, 59-61 months
  Distance between tantalum beads.
Time to Baseline Pain | Baseline, 2-6 weeks, 5-7 months, 11-13 months, 23-25 months, 59-61 months
  Visual Analog Scale
Quality of Life | Baseline, 2-6 weeks, 5-7 months, 11-13 months, 23-25 months, 59-61 months
  PROMIS Pain Interference and Mobility
Length of Hospital Stay | An expected average of 2 days
  participants will be followed for the duration of hospital stay (discharge date - admission date)
Time to full weight-bearing | 2- 6 weeks
  Documenting the number of days until patient could weight-bear without using devices as crutches or wheelchairs.
Need for Splint or Cast | 2- 6 weeks
  Documenting days worn.
Days Until Return to Sports | 2-6 weeks
  Documenting how many days elapsed before the patient returned to sports. This information will be recorded in a post-operative pain and function diary. Return to sports is typically surgeon driven, but timing for return to sports is not standardized in clinical practice. In the current study patients will be allowed to return to sports when pain free, no longer limping and strength is equivalent to the non-operative side
Need for Secondary Surgery | 2-6 weeks, 5-7 months, 11-13 months, 23-25 months, 59-61 months
  Assessed in follow up clinical visits and documented in clinical records
Physical Activity Level | Baseline, 2-6 weeks, 5-7 months, 11-13 months, 23-25 months, 59-61 months
  Pediatric activity scale assessment measured by HSS Pedi-FABS.
Physical Activity Level | Baseline, 2-6 weeks, 6 months, 12 months, 24 months, and 60 months
  UCLA Activity Scale
Complications | 2-6 weeks, 6 months, 12 months, 24 months, and 60 months
  Complications will be tracked for two years post surgery. Due to previous research, which is outlined below, the following complications will be included in the data collection follow up sheets: angular deformity, revision surgery, time until return to sports, hospital stay, failure/incomplete epiphysiodesis, time until weight bearing, infection, use of aid, number of days using the aid, and osteochondral damage.
Medical Costs | 5 years (end of study)
  Costs will be collected through hospital administration. In hospital costs and outpatients costs will be included. Indirect costs, such as lost days of parental work will not be considered. Only costs from the United States centers in this protocol will be assessed.
Operative Outcomes | intra-operative
  radiation, total time during surgery, skin dose, blood loss, surgeon experience, epiphysiodesis technique, fluoroscopy time
Radiographic Assessments | Baseline, 2-6 weeks, 5-7 months, 11-13 months, 23-25 months, 59-61 months
  Mechanical Tibial-Femoral Angle, Mechanical Axis Deviation, mLDFA, MPTA, PPTA

CONTACTS AND LOCATIONS:
Overall Officials: Emily R Dodwell, MD MPH FRCSC, Principal Investigator — Hospital for Special Surgery, New York
Locations (3):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Hospital for Special Surgery, New York, New York
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blair VP 3rd, Walker SJ, Sheridan JJ, Schoenecker PL. Epiphysiodesis: a problem of timing. J Pediatr Orthop. 1982 Aug;2(3):281-4. PMID 7130384
- [Background] Little DG, Nigo L, Aiona MD. Deficiencies of current methods for the timing of epiphysiodesis. J Pediatr Orthop. 1996 Mar-Apr;16(2):173-9. doi: 10.1097/00004694-199603000-00007. PMID 8742279
- [Background] Lauge-Pedersen H, Hagglund G, Johnsson R. Radiostereometric analysis for monitoring percutaneous physiodesis. A preliminary study. J Bone Joint Surg Br. 2006 Nov;88(11):1502-7. doi: 10.1302/0301-620X.88B11.17730. PMID 17075098
- [Background] Haugan K, Husby OS, Klaksvik J, Foss OA. The migration pattern of the Charnley femoral stem: a five-year follow-up RSA study in a well-functioning patient group. J Orthop Traumatol. 2012 Sep;13(3):137-43. doi: 10.1007/s10195-012-0187-x. Epub 2012 May 11. PMID 22576838
- [Background] Campens C, Mousny M, Docquier PL. Comparison of three surgical epiphysiodesis techniques for the treatment of lower limb length discrepancy. Acta Orthop Belg. 2010 Apr;76(2):226-32. PMID 20503949
- [Background] Ghanem I, Karam JA, Widmann RF. Surgical epiphysiodesis indications and techniques: update. Curr Opin Pediatr. 2011 Feb;23(1):53-9. doi: 10.1097/MOP.0b013e32834231b3. PMID 21169837
- [Background] DeWitt EM, Stucky BD, Thissen D, Irwin DE, Langer M, Varni JW, Lai JS, Yeatts KB, Dewalt DA. Construction of the eight-item patient-reported outcomes measurement information system pediatric physical function scales: built using item response theory. J Clin Epidemiol. 2011 Jul;64(7):794-804. doi: 10.1016/j.jclinepi.2010.10.012. Epub 2011 Feb 2. PMID 21292444
- [Background] Fabricant PD, Robles A, Downey-Zayas T, Do HT, Marx RG, Widmann RF, Green DW. Development and validation of a pediatric sports activity rating scale: the Hospital for Special Surgery Pediatric Functional Activity Brief Scale (HSS Pedi-FABS). Am J Sports Med. 2013 Oct;41(10):2421-9. doi: 10.1177/0363546513496548. Epub 2013 Jul 26. PMID 23893420
- [Background] Novais EN, Heyworth BE, Stamoulis C, Sullivan K, Millis MB, Kim YJ. Open surgical treatment of femoroacetabular impingement in adolescent athletes: preliminary report on improvement of physical activity level. J Pediatr Orthop. 2014 Apr-May;34(3):287-94. doi: 10.1097/BPO.0000000000000093. PMID 24172673
- [Background] Varni JW, Thissen D, Stucky BD, Liu Y, Magnus B, Quinn H, Irwin DE, DeWitt EM, Lai JS, Amtmann D, Gross HE, DeWalt DA. PROMIS(R) Parent Proxy Report Scales for children ages 5-7 years: an item response theory analysis of differential item functioning across age groups. Qual Life Res. 2014 Feb;23(1):349-61. doi: 10.1007/s11136-013-0439-0. Epub 2013 Jun 6. PMID 23740167
- [Background] Canale ST, Christian CA. Techniques for epiphysiodesis about the knee. Clin Orthop Relat Res. 1990 Jun;(255):81-5. PMID 2347169
- [Background] Metaizeau JP, Wong-Chung J, Bertrand H, Pasquier P. Percutaneous epiphysiodesis using transphyseal screws (PETS). J Pediatr Orthop. 1998 May-Jun;18(3):363-9. PMID 9600565
- [Background] Stewart D, Cheema A, Szalay EA. Dual 8-plate technique is not as effective as ablation for epiphysiodesis about the knee. J Pediatr Orthop. 2013 Dec;33(8):843-6. doi: 10.1097/BPO.0b013e3182a11d23. PMID 23872800
- [Background] Alzahrani AG, Behairy YM, Alhossan MH, Arab FS, Alammari AA. Percutaneous versus open epiphysiodesis. Saudi Med J. 2003 Feb;24(2):203-5. PMID 12682689